CLINICAL TRIAL: NCT02074306
Title: Does UROSHIELD® Influence Bacterial Growth On Endotracheal Tubes
Acronym: lungshield
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, REUVEN FRIEDMANN, head of geriatric ward, Shaare Zedek Medical Center
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 109/13; SZMCenter IRB (Other: Shaare Zedek Medical Center IRB)
Record Dates: First submitted 2014-02-13; First posted 2014-02-28 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Mechanical Ventilation Complication
Keywords: endotracheal intubation; low energy ultrasound; sputum culture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- UROSHIELD® (Experimental): Randomly selected patients,(ratio 1:1) with newly begun mechanical ventilation, will be connected to a low energy acustic wave generator UROSHIELD® within 48 hours. Endotracheal secretions will be collected for culture and antibiotic sensitivity every 3 days for 15 consecutive days or until disconnection from the mechanical ventilation.
  Interventions: Device: UROSHIELD®
- SHAM UROSHIELD® (Sham Comparator): same as abouve but with Sham device.
  Interventions: Device: SHAM UROSHIELD®

INTERVENTIONS:
Device: UROSHIELD® — An active UROSHIELD® device (low energy acustic wave generator) will be connected to an intratracheal tube externally. The device will transform low energy ultrasound waves on to the tube. These waves will by assumption lower the formation of bacterial growth and resistance to antibiotics.
  Other Names: LUNGSHIELD®
  Arms: UROSHIELD®
Device: SHAM UROSHIELD® — SHAM UROSHIELD® will be connected to endotracheal tubes unable to transform any waves.
  Other Names: SHAM LUNGSHIELD®
  Arms: SHAM UROSHIELD®

SUMMARY:
The purpose of this study is to examine the effect of UROSHIELD® (a device which generates low energy ultrasound waves) on development of bacterial colonies on endotracheal tubes, in patient receiving mechanical ventilation, and to determine whether this device lowers the rate of bacterial resistance to antibiotics.

DETAILED DESCRIPTION:
Ventilator Associated Pneumonia (VAP) is a common complication in patients treated by mechanical ventilation, supposedly related to development of bacterial colonization on the endotracheal tubes. Therefore many devices were designed to address this issue.

NanovibronixTM Company developed "UROSHIELD®" a device which generates low energy ultrasound wave in the nanometer range, and delivers these waves by an actuator which is connected externally to a urinary catheter. It was shown that using UROSHIELD®, there was reduction in development of bacterial colonies, and lower rate of resistance of bacteria to antibiotics.

Aim of the study:

To examine the effect of UROSHIELD® on development of bacterial colonies on endotracheal tubes, in patient receiving mechanical ventilation, and to determine whether this device lowers the rate of bacterial resistance to antibiotics.

Methods:

Consecutive patients, with newly begun mechanical ventilation, will be connected to UROSHIELD® within 48 hours. Endotracheal secretions will be collected for culture and antibiotic sensitivity every 3 days for 15 consecutive days or until disconnection from the mechanical ventilation. Half of the devices will be active for the study group; the other half will be sham for the control. The devices will externally look identical and will have a serial number which will remain secret.

Primary end point: The time to convert the sputum culture from negative to positive.

Secondary end points: The number of positive cultures with virulent bacteria and the rate of development of resistance to antibiotics will also be compared.

By statistical analysis the investigators conclude that enrollment of 33 patients into each group will allow significant results to be detected.

Should the study group show longer time to convert to positive bacterial culture and/or lower antibiotic resistance, the use of UROSHIELD®, should be examined in a larger study, with reduction of VAP as a primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients, with newly begun mechanical ventilation, will be connected to UROSHIELD® within 48 hours

Exclusion Criteria:

* Pediatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of days elapse until development of positive sputum culture | 15-20 days
  Sputum for culture will be obtained every 3 days. Number of days till sputum culture will convert from negative to positive one will be calculated and compared for the study and control groups.

SECONDARY OUTCOMES:
Type of bacteria and antibiotic sensitivity | 15-20 days
  Types of bacteria and their sensitivities to antibiotics will be evaluated. Comparison will be done between rate of growth of serious pathogens (e.g., Methicillin resistant staphylococcus aureus (MRSA),Vancomycin-Resistant Enterococci (VRE)) in the study and control groups.
  Rate of resistance development to antibiotics will also be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Friedmann, Dr, Study Director — Shaare Zedek Medical Center
Locations (1):
- Medical wing, Shaare Zedek Medical Center, Jerusalem, Israel